CLINICAL TRIAL: NCT01635673
Title: Effects of Whole Body Vibration Exercise on Metabolic Systems in Latino Boys
Acronym: VIBES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: VIBES
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2011-05

CONDITIONS: Effects of Whole Body Vibration Exercise on Metabolic Systems
Keywords: Exercise; Latino; Hispanic; Boys
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): A group that continues with their normal daily activities for the duration of the study
- Exercise Group (Experimental): This group exercises 3 times each week
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — Whole body vibration exercise 3 times per week
  Arms: Exercise Group

SUMMARY:
The purpose of this study is to determine if whole body vibration exercise improves insulin/glucose dynamics and bone metabolism in Latino Boys.

ELIGIBILITY:
Inclusion Criteria:

* Boy 8-10 years of age
* Tanner Stage I
* Age and gender BMI > 85th percentile
* Hispanic descent( all four grandparents of Hispanic descent)

Exclusion Criteria:

* Acute or chronic illness
* Any condition known to influence body composition, or insulin/glucose dynamics
* Musculoskeletal disease, injury, or orthopedic condition that would prevent exercise

Ages: 8 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Blood insulin | Baseline and week 10
  Change in basal insulin levels

SECONDARY OUTCOMES:
Bone Density | Baseline and week 10
  Change in bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schroeder, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC Biokinesiology and Physical Therapy, Clinical Exercise Research Center, Los Angeles, California, United States